CLINICAL TRIAL: NCT04678791
Title: To Investigate the Efficacy and Safety of Nimotuzumab Combined With Concurrent Chemoradiotherapy Versus Concurrent Chemoradiotherapy in the Treatment of Local Advanced Cervical Squamous Cell Carcinoma
Brief Title: Nimotuzumab Combined With Chemoradiotherapy Versus Chemoradiotherapy for Local Advanced Cervical Squamous Cell Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Junjie Wang, Principal Investigator, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M2020411
Record Dates: First submitted 2020-12-16; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Cervical Squamous Cell Carcinoma
MeSH Terms: interventions — nimotuzumab; Cisplatin; Brachytherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nimotuzumab+ chemoradiotherapy (Experimental): Patients receive nimotuzumab combined with cisplatin and undergo external-beam radiation and brachytherapy.
  Interventions: Drug: Nimotuzumab; Drug: Cisplatin; Radiation: External-beam radiation; Radiation: Brachytherapy
- Chemoradiotherapy (Active Comparator): Patients receive cisplatin and undergo external-beam radiation and brachytherapy
  Interventions: Drug: Cisplatin; Radiation: External-beam radiation; Radiation: Brachytherapy

INTERVENTIONS:
Drug: Nimotuzumab — Patients receive Nimotuzumab 400 mg each time, once a week, slow intravenous drip, for a total of 6 weeks.
  Other Names: EGFR monoclonal antibody
  Arms: Nimotuzumab+ chemoradiotherapy
Drug: Cisplatin — Patients receive 40 mg/m2, d1, 7 days as 1 treatment cycle, 6 treatment cycles in total
  Other Names: Cisplatin injection
Radiation: External-beam radiation — Patients undergo IMRT/VMAT radiotherapy with pelvic and/or extended field irradiation at a total dose of 45 - 50.4 Gy; 1.8 - 2.0 Gy/f, 25 - 28 f.
Radiation: Brachytherapy — Patient undergo Brachytherapy with high dose rate, with a total dose of 30-40 Gy and a cumulative dose of 80 ~ 85 Gy at point A/HRCTV D90; if the tumor diameter is ≥ 4 cm, the cumulative dose of ≥ 87 Gy at point A/HRCTV D90.

SUMMARY:
To investigate the efficacy and safety of nimotuzumab combined with concurrent chemoradiotherapy versus concurrent chemoradiotherapy in the treatment of local advanced cervical squamous cell carcinoma.

DETAILED DESCRIPTION:
This study adopts a multi-center, randomized controlled, open-label clinical trial design.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years old;
2. Histologically diagnosed primary cervical squamous cell carcinoma, with clinical stage IB3-IVA (FIGO 2018);
3. At least one measurable lesion according to RECIST 1.1;
4. Absence of severe hematopoietic dysfunction and heart, lung, liver, kidney dysfunction and immunodeficiency, laboratory test results meet the following criteria:

   Hemoglobin ≥ 90 g/L; Absolute neutrophil count ≥ 2 × 109/L or white blood cell count ≥ 4.0 × 109/L; Platelet count ≥ 100 × 109/L; Aspartate aminotransferase (AST) ≤ 2.5 × ULN Alanine aminotransferase (ALT) ≤ 2.5 × ULN Total bilirubin ≤ 1.5 × ULN; Serum creatinine ≤ 1.0 × ULN;
5. ECOG score 0-2 points;
6. Expected survival ≥ 3 months;
7. Women of childbearing potential must have a negative serum or urine HCG within 72 hours prior to enrollment (postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential. A pregnancy test is not required for women who have demonstrated tubal ligation);
8. No intrauterine device;
9. Women of childbearing potential who are willing to take medically recognized contraceptive measures during the trial;
10. Compliance is good and informed consent is voluntarily signed.

Exclusion Criteria:

1. Cervical adenocarcinoma and rare pathological types of malignant tumors;
2. Previous surgery for cervical cancer, pelvic radiation therapy, systemic chemotherapy, tumor targeted therapy, immunotherapy;
3. Ureteral obstruction, inability to place ureteral stent or pyelostomy;
4. Pregnant or lactating women;
5. Patients with rectovaginal fistula/vaginovesical fistula/uncontrolled vaginal bleeding or at risk of fistula;
6. Human immunodeficiency virus (HIV) infection;
7. Active hepatitis B (the quantitative detection result of HBV DNA exceeds the lower limit of detection), or HCV infection (the quantitative detection result of HCV RNA exceeds the lower limit of detection);
8. Patients have a serious underlying condition that precludes safe administration of trial treatment. Including but not limited to active infection requiring systemic drug therapy: decompensated heart failure (NYHA Class III and IV), unstable angina pectoris, acute myocardial infarction within 3 months prior to enrollment;
9. Patients with a history of other malignant tumors (except cured cutaneous basal cell carcinoma);
10. Patients with Crohn's disease and ulcerative colitis;
11. Patients who are participating in other clinical trials or have stopped clinical trials for less than 4 weeks;
12. Patients with known hypersensitivity to Nimotuzumab or its components;
13. Patients with contraindications to cisplatin;
14. Patients with neurological or psychiatric disorders affecting cognitive ability;
15. Patients whose lesions cannot be treated with intracavitary radiotherapy as assessed by the investigator;
16. Other reasons that, in the judgment of the investigator, would make the patient inappropriate for the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
3-year progression-free survival (PFS) | up to 3 years
  The rate of patient without progress disease in 3 years after treatment

SECONDARY OUTCOMES:
3-year overall survival (OS) | up to 3 years
  The rate of patient alive in 3 years after treatment
Complete response rate (CRR) | 3 months later after treatment
  Percentage of subjects in this group who achieve complete response by imaging assessment from the end of treatment to disease progression.
Objective response rate (ORR) | 3 months later after treatment
  The percentage of patients who experienced complete or partial cancer shrinkage or disappearance after treatment.
Incidence and severity of acute adverse events | up to 3 months complete treatment
  Number and grade of participants with adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University 3rd Hospital, Beijing, Beijng, China

IPD SHARING:
Plan to Share IPD: No